CLINICAL TRIAL: NCT04787549
Title: Effect of Cognitively Challenging Exergames Using Fully Immersive Virtual Reality in Patients With Parkinson's Disease: A Pilot Study
Brief Title: Effect of Immersive Virtual Reality Exergames in Patients With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Han Gil Seo, Associate Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PD-VR-pilot
Record Dates: First submitted 2021-03-01; First posted 2021-03-08 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; Virtual reality; Exergame
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual reality exergames (Experimental): Cognitively challenging exergames using fully immersive virtual reality with a head-mounted display (HTC Vive; HTC Co., New Taipei City, Taiwan)
  Interventions: Device: Virtual reality exergames

INTERVENTIONS:
Device: Virtual reality exergames — A total of 10 sessions were held for 30 minutes, 2 to 3 times a week for exergames using fully immersive virtual reality under the assistance of an occupational therapist.

SUMMARY:
The study aimed to investigate the effect of applying cognitively challenging exergames using fully immersive virtual reality in patients with Parkinson's disease.

DETAILED DESCRIPTION:
It has been reported that dual-task training involving both cognitive and physical functions helps improve walking speed during dual-task performance without increasing the fall risk in patients with Parkinson's disease (PD). Compared with conventional physical therapy, there are studies that dual-task training significantly improved walking speed and stride in PD patients. In addition, a systematic review study has been reported that it helps to improve balance and cognitive function when dual-task training is performed for patients with neurological diseases including Parkinson's disease.

Virtual reality is expected to promote functional recovery in patients with neurological disorders in terms of providing an enriched environment, goal-directed tasks and repetition, and inducing interest and motivation. Therefore, the study aimed to investigate the effect of applying cognitively challenging exergames using fully immersive virtual reality in patients with PD.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed as idiopathic Parkinson's disease
* Modified Hoehn & Yahr stage 2, 2.5, or 3

Exclusion Criteria:

* Moderate to severe cognitive dysfunction with Mini-mental State Examination score < 19
* Severe dyskinesia or severe on-off phenomenon
* Plan to adjust medication at the time of screening
* Other brain diseases such as stroke, brain tumor, etc
* History of seizure
* Vestibular disease or paroxysmal vertigo
* Other comorbidities that make it difficult to participate in this study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2022-01-27 (Actual); Study Completion 2022-01-27 (Actual)

PRIMARY OUTCOMES:
Cognitive dual-task interference (%) in Timed-up & go test | at study completion, an average of 1 month
Physical dual-task interference (%) in Timed-up & go test | at study completion, an average of 1 month

SECONDARY OUTCOMES:
Timed-up & go test (sec): single task | at study completion, an average of 1 month
Timed-up & go test (sec): cognitive dual-task | at study completion, an average of 1 month
Timed-up & go test (sec): physical dual-task | at study completion, an average of 1 month
The Unified Parkinson's Disease Rating Scale | at study completion, an average of 1 month
  The higher the score, the more negative the result
Berg balance scale | at study completion, an average of 1 month
  The higher the score, the more positive the result
Stroop test | at study completion, an average of 1 month
Trail making test | at study completion, an average of 1 month
Digit span test | at study completion, an average of 1 month
New Freezing of Gait Questionnaire (NFOGQ) | at study completion, an average of 1 month

OTHER OUTCOMES:
Simulator sickness questionnaire (SSQ) | at 1st session (an average of 3 days) and at study completion (an average of 1 month)

CONTACTS AND LOCATIONS:
Overall Officials: Han Gil Seo, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Yun SJ, Hyun SE, Oh BM, Seo HG. Fully immersive virtual reality exergames with dual-task components for patients with Parkinson's disease: a feasibility study. J Neuroeng Rehabil. 2023 Jul 18;20(1):92. doi: 10.1186/s12984-023-01215-7. PMID 37464349